CLINICAL TRIAL: NCT02368093
Title: A Double-blind, Placebo-controlled, Therapeutic Trial With Antitussive Drug-Dextromethorphan: Aimed to Determine Its Therapeutic Effect in Patients With Rheumatoid Arthritis
Brief Title: Efficacy Study of Dextromethorphan to Treat Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C09060-1
Record Dates: First submitted 2015-02-04; First posted 2015-02-20 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dextromethorphan hydrobromide (Experimental): Dextromethorphan hydrobromide; Detosiv Slow Release® (60mg per tablet, Lotus Pharmaceutical Company, Taipei, Taiwan), 120mg per day with once daily dose taken after breakfast]
  Interventions: Drug: Dextromethorphan hydrobromide
- Placebo (Placebo Comparator): placebo pills with the same appearance as Detosiv tablets.

INTERVENTIONS:
Drug: Dextromethorphan hydrobromide — 120mg per day with once daily dose taken after breakfast for 6 months
  Other Names: Detosiv Slow Release®
  Arms: Dextromethorphan hydrobromide

SUMMARY:
Rheumatoid arthritis were randomized to a 6-month treatment of oral dextromethorphan hydrobromide or placebo as an add-on therapy to traditional disease-modifying anti-rheumatic drugs (DMARDs). Disease activity were assessed.

DETAILED DESCRIPTION:
Biologic-naïve rheumatoid arthritis (RA) patients who fulfilled the 2010 criteria of the American College of Rheumatology (ACR) for RA were enrolled. All patient were randomized to a 6-month treatment with either oral DXM [dextromethorphan hydrobromide; Detosiv Slow Release® (60mg per tablet, Lotus Pharmaceutical Company, Taipei, Taiwan) with T1/2 = 7.75h, Tmax = 4.83h, Cmax = 14.6 ng mL-1 and mean residual time = 5.86 h, 120mg per day with once daily dose taken after breakfast] or placebo pills with the same appearance as DXM tablets. The randomization was performed by the pharmacy of the Taichung Veterans General Hospital. Non-study medications were not changed during the course of study.

Twenty-four patients received add-one DXM therapy and the other 24 patients received traditional DMARDs alone in stable dose. Disease activity was assessed by the 28-joint disease activity score (DAS28) before starting add-on DXM therapy (as a baseline) and at the end of 6 months of therapy with or without add-on DXM. Patients were categorized as good, moderate or poor responders based on the amount of change in the DAS28 and the level of DAS28 reached. Good responders were defined as patients who had a decrease in DAS28 from baseline (∆DAS28)>1.2 and a DAS28≦3.2 at evaluation time; moderate responders had either ∆DAS28>1.2 and a DAS28>3.2 or ∆DAS28 of 0.6-1.2 and a DAS28≦5.1 at evaluation time; and poor responders were those who had either ∆DAS28<0.6 or a DAS28>5.1 at evaluation time.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the 2010 criteria of the American College of Rheumatology (ACR) for RA

Exclusion Criteria:

* Receive biological therapy for RA, including Etanercept, Adalimumab, Golimumab, Tocilizumab, Rituximab, Abatacept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Der-Yuan Chen, M.D., Ph.D., Principal Investigator — Division of Allergy,Immunology and Rheumatology, Taichung Veterans General Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Dextromethorphan: Biologic-naïve rheumatoid arthritis patients who fulfilled the 2010 criteria of the American College of Rheumatology for RA were enrolled.
  Dextromethorphan hydrobromide 120mg once daily were given for 6 months.
- Placebo: Biologic-naïve rheumatoid arthritis patients who fulfilled the 2010 criteria of the American College of Rheumatology for RA were enrolled.
  Placebo pills with the same appearance as Dextromethorphan hydrobromide tablets once daily were given for 6 months.
Period: Overall Study
Arm/Group | Dextromethorphan | Placebo
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dextromethorphan Hydrobromide: Dextromethorphan hydrobromide; Detosiv Slow Release® (60mg per tablet, Lotus Pharmaceutical Company, Taipei, Taiwan), 120mg per day with once daily dose taken after breakfast for 6 months
- Placebo: Placebo pills with the same appearance as Detosiv tablets once daily for 6 months.
- Total: Total of all reporting groups
Arm/Group | Dextromethorphan Hydrobromide | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.6) | 52.8 (10.5) | 52.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants] — Ethnicity of participants
  participants
    Taiwan | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Good European League Against Rheumatism (EULAR) Therapeutic Response Rate
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 24 | 24
participants | 6 | 4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dextromethorphan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No